CLINICAL TRIAL: NCT04787965
Title: Opicapone Treatment Initiation Open-Label Study
Acronym: OPTI-ON
Status: Completed | Type: Observational
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: NBI-OPC-PD4006
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease (PD); Levodopa; Carbidopa; Motor Fluctuations; Non-Motor Fluctuations; Adjunctive treatment; COMT inhibitor
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ONGENTYS: Opicapone 50 mg capsule once daily for 6 months
  Interventions: Drug: Opicapone

INTERVENTIONS:
Drug: Opicapone — Opicapone as adjunctive treatment to levodopa/carbidopa over a 6-month period
  Other Names: ONGENTYS

SUMMARY:
This is an observational study to describe the treatment patterns and clinical outcomes observed with use of ONGENTYS as adjunctive treatment to levodopa/carbidopa in Parkinson's disease patients experiencing "off" episodes with motor fluctuations

ELIGIBILITY:
Inclusion Criteria:

* Must be able to complete electronic patient-reported outcome instruments
* Parkinson's disease patients experiencing "off" episodes
* Patient receiving concomitant levodopa/carbidopa, and as deemed appropriate by the physician, newly initiating ONGENTYS as adjunctive treatment

Exclusion Criteria:

* Patient is not cognitively able to complete the study requirements
* Patient is not able to complete the study duration of 6 months
* History of moderate or severe hepatic impairment
* Patient has end-stage renal disease
* Concomitant use of non-selective monoamine oxidase (MAO) inhibitor or catechol-O-methyltransferase (COMT) inhibitors (patients entering study may switch from other COMT inhibitors to ONGENTYS)
* History of pheochromocytoma, paraganglioma, or other catecholamine-secreting neoplasms
* Currently enrolled in an interventional clinical trial
* Currently or previously received ONGENTYS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients experiencing "off" episodes with motor fluctuations, who are currently being treated by a neurologist and require adjunctive treatment to levodopa/carbidopa
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
ONGENTYS treatment patterns | 6 months
  Reason for initiating treatment and discontinuation

SECONDARY OUTCOMES:
PD Status | 6 months
  PD Status Questionnaire
CGI-C | 6 months
  Clinical Global Impression of Change Scale
MDS-UPDRS Parts I, II, and IV | 6 months
  Movement Disorder Society-Unified Parkinson's Disease Rating Scale
PDQ-8 | 6 months
  Parkinson's Disease Questionnaire-8
PGI-C | 6 months
  Patient Global Impression of Change Scale
NoMoFa | 6 months
  Non-Motor Fluctuation Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Olga Klepitskaya, MD, FAAN, Study Director — Neurocrine Biosciences
Locations (6):
- United States (6):
  - Neurocrine clinical site, Los Gatos, California
  - Neurocrine clinical site, Memphis, Tennessee
  - Neurocrine clinical site, Christiansburg, Virginia
  - Neurocrine clinical site, Norfolk, Virginia
  - Neurocrine clinical site, Auburn, Washington
  - Neurocrine clinical site, Crab Orchard, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferreira JJ, Lees A, Rocha JF, Poewe W, Rascol O, Soares-da-Silva P; Bi-Park 1 investigators. Opicapone as an adjunct to levodopa in patients with Parkinson's disease and end-of-dose motor fluctuations: a randomised, double-blind, controlled trial. Lancet Neurol. 2016 Feb;15(2):154-165. doi: 10.1016/S1474-4422(15)00336-1. Epub 2015 Dec 23. PMID 26725544
- [Background] Lees AJ, Ferreira J, Rascol O, Poewe W, Rocha JF, McCrory M, Soares-da-Silva P; BIPARK-2 Study Investigators. Opicapone as Adjunct to Levodopa Therapy in Patients With Parkinson Disease and Motor Fluctuations: A Randomized Clinical Trial. JAMA Neurol. 2017 Feb 1;74(2):197-206. doi: 10.1001/jamaneurol.2016.4703. PMID 28027332